CLINICAL TRIAL: NCT05934032
Title: Registry of the National Network Genomic Medicine Lung Cancer (nNGM), Linking Data on Molecular Diagnostics, Clinical Characteristics, Treatment Patterns and Outcomes of Subjects With Non-Small Cell Lung Cancer in Germany
Brief Title: National Network Genomic Medicine Lung Cancer, Germany
Acronym: nNGM
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Juergen Wolf (Other)
Collaborators: Charite University, Berlin, Germany (Other); Helios Klinikum Emil von Behring (Unknown); Vivantes Hospital Berlin Neukölln (Unknown); University Hospital Carl Gustav Carus (Other); Heinrich-Heine University, Duesseldorf (Other); University Hospital Erlangen (Other); University Hospital, Essen (Other); Goethe University (Other); University Hospital Freiburg (Other); University Hospital Giessen and Marburg (Unknown); University Hospital Halle (Saale) (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Heidelberg (Other); Klinikum Hanover-Siloah Hospital (Other); University Hospital, Bonn (Other); University Hospital Schleswig-Holstein (Other); Johannes Gutenberg University Mainz (Other); University Hospital Munich (LMU) (Unknown); University Hospital rechts der Isar Munich (TUM) (Unknown); Pius-Hospital Oldenburg (Other); University Hospital Regensburg (Other); University Hospital Tuebingen (Other); Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); University Hospital Ulm (Other); Wuerzburg University Hospital (Other); University Hospital of Cologne (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Juergen Wolf, Professor Dr. med., Spokesperson of the National Network Genomic Medicine Lung Cancer, University of Cologne
Organization: University of Cologne (Other)
Other Study IDs: NNGM0418
Record Dates: First submitted 2023-06-16; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: carcinoma, non-small-cell lung* / diagnosis; carcinoma, non-small-cell lung* / genetics; precision medicine; lung neoplasms; neoplasms by site; registry; pathology, molecular
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Disease; Lung Neoplasms; Neoplasms by Site

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational, non-interventional — observational, non-interventional

SUMMARY:
Registry of the national Network Genomic Medicine Lung Cancer (nNGM), linking data on molecular diagnostics, clinical characteristics, treatment patterns and outcomes of subjects with non-small cell lung cancer (NSCLC) from 23 specialized cancer centres and more than 400 general hospitals and oncological practices in Germany

DETAILED DESCRIPTION:
Within the national Network Genomic Medicine Lung Cancer (nNGM), comprehensive molecular diagnostics and treatment recommendations are provided by 23 certified cancer centres according to standardized procedures for patients with non-resectable NSCLC. More than 400 network partners across Germany (including hospitals and oncological practices) report data on subsequent treatment and outcomes to the nNGM registry. Clinical outcomes are continuously evaluated through analysis of data collected in a decentralized registry. The nNGM registry records the patient journey and course of the disease from first histologically confirmed diagnosis to death or loss to follow-up and comprises detailed data on demographic and clinical characteristics, molecular diagnostics (including comprehensive biomarker testing results), treatments (targeted therapy, immunotherapy, chemotherapy, radiotherapy, best supportive care) and outcomes (overall survival, response, disease progression, time to next treatment). Patients have been actively involved throughout all stages of the design and running of the network and its registry.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed, locally advanced or metastatic NSCLC (Union for International Cancer Control [UICC] stage IIIb/IV; non-resectable NSCLC)
* From 07/2023: histologically confirmed NSCLC stage Ib, II, III (UICC)

Exclusion Criteria:

* Missing written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with histologically confirmed NSCLC are enrolled by 23 certified cancer centres and more than 400 network partners (hospitals and oncological practices) across Germany.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
molecular testing | 1 year
  descriptive data on results, frequency and methods of molecular testing
treatment patterns | from first diagnosis to death or loss to follow-up, whichever came first, assessed up to 100 months
  descriptive data on systemic treatments (including combination and sequence of treatments)
overall survival | assessed up to 100 months
  overall survival (in months)
time to next treatment | from start of treatment to the start of the next therapy, death or loss to follow-up, whichever came first, assessed up to 100 months
  time to next treatment (in months)
progression free survival | from start of treatment to tumour progression, death or loss to follow-up, whichever came first, assessed up to 100 months
  progression free survival (in months)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Wolf, Prof. Dr., Study Chair — University of Cologne
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Janning M, Suptitz J, Albers-Leischner C, Delpy P, Tufman A, Velthaus-Rusik JL, Reck M, Jung A, Kauffmann-Guerrero D, Bonzheim I, Brandlein S, Hummel HD, Wiesweg M, Schildhaus HU, Stratmann JA, Sebastian M, Alt J, Buth J, Esposito I, Berger J, Togel L, Saalfeld FC, Wermke M, Merkelbach-Bruse S, Hillmer AM, Klauschen F, Bokemeyer C, Buettner R, Wolf J, Loges S; National Network Genomic Medicine Lung Cancer (nNGM). Treatment outcome of atypical EGFR mutations in the German National Network Genomic Medicine Lung Cancer (nNGM). Ann Oncol. 2022 Jun;33(6):602-615. doi: 10.1016/j.annonc.2022.02.225. Epub 2022 Mar 6. PMID 35263633
- [Background] Saleh MM, Scheffler M, Merkelbach-Bruse S, Scheel AH, Ulmer B, Wolf J, Buettner R. Comprehensive Analysis of TP53 and KEAP1 Mutations and Their Impact on Survival in Localized- and Advanced-Stage NSCLC. J Thorac Oncol. 2022 Jan;17(1):76-88. doi: 10.1016/j.jtho.2021.08.764. Epub 2021 Sep 30. PMID 34601169
- [Background] Saalfeld FC, Wenzel C, Christopoulos P, Merkelbach-Bruse S, Reissig TM, Lassmann S, Thiel S, Stratmann JA, Marienfeld R, Berger J, Desuki A, Velthaus JL, Kauffmann-Guerrero D, Stenzinger A, Michels S, Herold T, Kramer M, Herold S, Tufman A, Loges S, Alt J, Joosten M, Schmidtke-Schrezenmeier G, Sebastian M, Stephan-Falkenau S, Waller CF, Wiesweg M, Wolf J, Thomas M, Aust DE, Wermke M; National Network Genomic Medicine Lung Cancer (nNGM). Efficacy of Immune Checkpoint Inhibitors Alone or in Combination With Chemotherapy in NSCLC Harboring ERBB2 Mutations. J Thorac Oncol. 2021 Nov;16(11):1952-1958. doi: 10.1016/j.jtho.2021.06.025. Epub 2021 Jul 8. PMID 34245914
- See also: Website of the national Network Genomic Medicine Lung Cancer, Germany — https://nngm.de